CLINICAL TRIAL: NCT01254474
Title: Evaluation of Depolarization and Repolarisation Activity During Cardiac Arrhythmia Using a Novel Monophasic Action Potential Catheter
Acronym: EvaMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2010/42
Record Dates: First submitted 2010-12-01; First posted 2010-12-06 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation; Ventricular Fibrillation; Junctional Tachycardia
Keywords: Depolarization, tissue; Repolarization, tissue; Cardiac Arrhythmias; Action potentials, monophasic; Mapping, Catheter; Cardiac activation
MeSH Terms: conditions — Atrial Fibrillation; Ventricular Fibrillation; Tachycardia, Ectopic Junctional; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MAP 4 procedure (Experimental): Assess MAP 4 mapping capabilities in cardiac chambers in patients suffering from regular or fibrillating tachycardia's
  Interventions: Device: Cardiac chambers mapping with MAP 4

INTERVENTIONS:
Device: Cardiac chambers mapping with MAP 4

SUMMARY:
Monophasic action potential (MAP) recording plays an important role in a more direct view of human myocardial electrophysiology under both physiological and pathological conditions. The MAP method represents a very useful tool for an electrophysiological research in cardiology. Its crucial importance lies in the fact that it enables the study of the action potential (AP) of myocardial cell in vivo and, therefore, the study of the dynamic relation of this potential with all the organism variables what can be particularly helpful in the case of arrhythmias.

Hundred and fifty patients will be included to explore mapping capabilities in cardiac chambers in patients suffering from regular or fibrillating tachycardia's with the following inclusion plan: i) Atrial fibrillation at a total of 50 patients ii) Ventricular fibrillation or patients at high risk of sudden cardiac death at a total of 50 patients iii) Junctional tachycardia at a total of 50 patients. We will focus on cardiac activation (depolarization and repolarization) in this population.

DETAILED DESCRIPTION:
This is a prospective descriptive study including 1 French centre The arrhythmogenic substrate that leads to fibrillating heart is poorly understood. This has hindered the development of methods for better understanding mechanisms. The development of better adapted tools to improve understanding and assessment of this substrate is crucial. The current electrophysiological study preceding the ablation is exclusively based on substrate depolarisation potential. It is very powerful when the arrhythmia is organized but limited during fibrillation due to incessant changes in activation. Therefore, potentials of repolarization are better suited for the explorations of fibrillations because they provide basic properties such as refractory period and tissue heterogeneity in arrhythmia, but also in sinus rhythm. Monophasic Action Potential catheters (MAP EFA Boston and MAP Biosense Webster) are available for many years and represent a very useful tool in cardiology in identifying critical areas to arrhythmias (mapping of depolarization and cardiac repolarization). However, their capacity to record action potential is limited because they have one electrode that allows "point-to-point" mapping by moving the catheter sequentially in the cardiac cavities. Moreover, it is difficult to obtain one action potential due to the configuration or the angle of contact of the catheter with the cardiac wall. We want to evaluate a new MAP catheter (MAP4, Medtronic) to assess cardiac depolarization and repolarization. This catheter was developed to allow recording of an action potential whenever the catheter touches the heart wall and whatever the configuration or contact angle. It appears identical to other catheters but is equipped with 4 spherical microelectrodes at its end. Each microelectrode is arranged to one of the 4 'cardinal points' which allows easily simultaneous recording of 4 actions potential. Hundred and fifty patients will be included to explore mapping capabilities in cardiac chambers in patients suffering from regular or fibrillating tachycardia's with the following inclusion plan: i) Atrial fibrillation at a total of 50 patients ii) Ventricular fibrillation or patients at high risk of sudden cardiac death at a total of 50 patients iii) Junctional tachycardia at a total of 50 patients. We will focus on cardiac activation (depolarization and repolarization) in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atrial Fibrillation or Ventricular Fibrillation or junctional tachycardia or reentrant tachycardia
* Age ≥ 18 years old
* Signed patient informed consent form
* Affiliated to social security (European countries)

Exclusion Criteria:

* Patients under 18 years old
* Pregnancy
* Psychiatric disorders
* Neurological sequelae after a prior cardiac arrest that prevents informed consent
* Absence of informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-04-12 (Actual)

PRIMARY OUTCOMES:
Cardiac activation identified during the intervention by depolarization and repolarization times | End of mapping procedure (up to 5 days after inclusion)
  The performance criteria of this MAP4 catheter will be evaluated in providing information on the action potentials to further improve insight into mechanisms.
  Cardiac activation (depolarization and repolarization) identified during the intervention with established criteria:
  * abnormal depolarization will be defined by a local delay of conduction >25 ms.
  * abnormal repolarization will be defined if a gradient of repolarization > 50 ms.

SECONDARY OUTCOMES:
Presence of zone of low voltage (<0.5 mV) | End of mapping procedure (up to 5 days after inclusion)
Presence of post depolarization on MAP4 catheter | End of mapping procedure (up to 5 days after inclusion)
Adverse events during procedure and/or during 6 months | 6 months
Skin to skin procedural time | End of mapping procedure (up to 5 days after inclusion)
  Skin to skin procedural time (major reduction of time mapping is expected with MAP4. This variable is appreciated by the duration of the procedure and fluoroscopic time (in minutes))

CONTACTS AND LOCATIONS:
Overall Officials: Mélèze HOCINI, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Hôpital cardiologique du Haut-Lévêque, Cardiac arrhythmias department, Pessac, France